CLINICAL TRIAL: NCT02451735
Title: Genetic Counseling for Breast Cancer Survivors (GC for BC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-16723
Record Dates: First submitted 2015-05-18; First posted 2015-05-22 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: female breast cancer; bilateral breast cancer; triple negative breast cancer; breast cancer diagnosis; BRCA 1; BRCA 2; psychoeducational intervention (PEI); genetic counseling; hereditary breast and ovarian cancer (HBOC); cancer education materials
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Development (No Intervention): Psychoeducational Intervention (PEI) development. PEIs include printed and DVD materials, and represent a commonly used and effective approach to implement theoretically based individual-level interventions. These materials serve as important sources of information for the general public, cancer patients, and survivors from a variety of backgrounds, including populations with limited health literacy. An interview and feedback collection process will take place to provide data to improve current PEI materials.
- Intervention Pilot - Intervention Group (Experimental): The intervention group will receive the PEI materials: video and booklet. Self-reported feedback will be collected and reviewed to compare response with the control group.
  Interventions: Behavioral: Video and Booklet
- Intervention Pilot - Control Group (Active Comparator): The control group will receive a patient factsheet about Genetic Counseling (GC). Self-reported feedback will be collected and reviewed to compare response with the intervention group.
  Interventions: Behavioral: Factsheet

INTERVENTIONS:
Behavioral: Video and Booklet — Printed and DVD materials about Genetic Counseling. Self-reported feedback will be collected and reviewed to compare to the control group response.
  Arms: Intervention Pilot - Intervention Group
Behavioral: Factsheet — Patient factsheet about Genetic Counseling. Self-reported feedback will be collected and reviewed to compare to the intervention group response.
  Arms: Intervention Pilot - Control Group

SUMMARY:
The purpose of this study is to review and evaluate the effectiveness of new educational materials (informational booklet & DVD) that promote participation in genetic counseling among breast cancer survivors.

There are two phases to this study:

Part 1 - reviewing the newly developed educational materials, and Part 2 - evaluating the effectiveness of the newly developed educational materials

DETAILED DESCRIPTION:
Part 1: Intervention Development

Aim 1: Develop a psychoeducational intervention (PEI) for high-risk breast cancer survivors about genetic counseling (GC) and hereditary breast and ovarian cancer (HBOC).

Part 2: Intervention Pilot

Aim 2: Assess the feasibility and acceptability of a PEI from the perspective of the BC patients and health care professionals.

Exploratory Aim 3: Estimate the preliminary efficacy of the PEI compared to standard clinical care. We hypothesize that women in the intervention group will have higher uptake of GC, greater increases in knowledge, and more perceived benefits related to GC compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

Part 1: Female breast cancer patients at Moffitt Cancer Center (MCC) are eligible to participate if they:

* are > 18 years of age;
* have no documented or observable psychiatric or neurological disorders that would interfere with study participation (e.g., dementia, psychosis);
* are capable of speaking and reading standard English;
* have not attended or scheduled an upcoming appointment for genetic counseling at the time of recruitment;
* are within 18 months of their breast cancer (BC) diagnosis;
* have a previous diagnosis of breast cancer or;
* received a referral letter for GC from their MCC physician;
* breast cancer at age 50 or below;
* bilateral breast cancer;
* multiple cancers except basal cell carcinoma;
* triple negative breast cancer;
* ovarian cancer or fallopian tube cancer at any age;
* of Ashkenazi Jewish descent;
* have 2 or more blood relatives diagnosed with breast cancer;
* have any blood relatives diagnosed with bilateral breast cancer;
* a first degree relative diagnosed with breast cancer below age 50;
* have blood relatives diagnosed with ovarian cancer;
* have 2 or more family members on the same side of the family with breast, ovarian, pancreatic, or prostate cancer;
* have a known cancer gene mutation (such as BRCA 1/2;
* have any male relatives diagnosed with breast cancer ; and
* have a mailing address and working telephone number; and
* provide written informed consent.

Part 2: Female BC patients at MCC are eligible to participate if they:

* are > 18 years of age;
* have no documented or observable psychiatric or neurological disorders that would interfere with study participation (e.g., dementia, psychosis);
* are capable of speaking and reading standard English;
* have not attended or scheduled an upcoming appointment for GC at the time of recruitment;
* have a previous diagnosis of breast cancer or;
* received a referral letter for GC from their MCC physician;
* breast cancer at age 50 or below;
* bilateral breast cancer;
* multiple cancers except basal cell carcinoma;
* triple negative breast cancer;
* ovarian cancer or fallopian tube cancer at any age
* of Ashkenazi Jewish descent;
* have 2 or more blood relatives diagnosed with breast cancer;
* have any blood relatives diagnosed with bilateral breast cancer;
* a first degree relative diagnosed with breast cancer below age 50;
* have blood relatives diagnosed with ovarian cancer;
* have 2 or more family members on the same side of the family with breast, ovarian, pancreatic, or prostate cancer;
* have a known cancer gene mutation (such as BRCA 1/2;
* have any male relatives diagnosed with breast cancer ; and
* have a mailing address and working telephone number; and
* provide written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2012-07-27 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Part 1: Rate of Initial Survey Responses | Up to 8 months
  Intervention Development: Rate of feedback of draft materials required to complete a formative evaluation.
Part 2: Rate of Participation | Up to 8 months
  Participation in the Psychoeducational Intervention (PEI) group compared to the Factsheet group.

SECONDARY OUTCOMES:
Rate of Impact | Up to 8 months
  Self-Reported Feedback Scoring Method: Frequencies and descriptives will be calculated for response options. Positive feedback rate of Psychoeducational Intervention (PEI) group compared to the Factsheet group.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Vadaparampil, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States